CLINICAL TRIAL: NCT04698811
Title: Virtual Eneagram: Quality of Life, Stress and Anxiety.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, José Dias da Silva Neto, Director, Universidade do Vale do Sapucai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Fundação de Ensino Superior
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Personality
Keywords: Personality. .; Anxiety; Quality of Life.; Stress, Psychological.; Personality Tests.
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be invited to the activities through the publication of registration on social networks. After reading and accepting the informed consent form, the initial information for the design of the group will be filled out. The activities will be applied to a minimum group of 135 people. If the number of registrants qualified for the study does not reach 135 individuals, the registration period will be extended by 15 days in order to complete the sample. Still being insufficient, the test will be carried out with the sample found.
Masking Description: Masking will not occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIRTUAL ENEAGRAM: QUALITY OF LIFE, STRESS AND ANXIETY. (Other): Training and testing battery.
  Interventions: Behavioral: VIRTUAL ENEAGRAM

INTERVENTIONS:
Behavioral: VIRTUAL ENEAGRAM — Presentation of the Virtual Enneagram and its content and realization of the first battery of tests (World Health Organization Quality of Life - (WHOQOL-BREF). Stress Perception Scale 10 (EPS-10) The Trait-State Anxiety Inventory: IDATE E and T.) .
  Guidance and training on personality and the Enneagram, its classification system, personality subtypes and dynamics of stress and growth allowing self-recognition.
  Second test battery ((World Health Organization Quality of Life - (WHOQOL-BREF). Stress Perception Scale 10 (EPS-10) The Trait-State Anxiety Inventory: (IDATE E and T.) and Enneagram Questionnaire.

SUMMARY:
The objetictive is to observe the influence of the enneagram typology on the perception of anxiety, stress and quality of life through self-knowledge directed in a virtual learning environment. The study is a clinical, primary, analytical, prospective and longitudinal study. It will be carried out in a virtual learning environment (VLE) with the collection of data obtained before and after the beginning of the training on the enneagram. The training will be divided into three online AVA modules. Casuistry: after orientations and signature of the term (Informed Consent Form), they will register on social networks where the initial information will be filled out. to outline the group. Inclusion criteria: participants of both sexes, Brazilians, over 18 years old; agree to sign the Informed Consent Form; with the desire to realize self-knowledge with the availability of time and access to the internet to hold meetings; Non-inclusion criteria: do not have previous information about the enneagram and speak the Portuguese language; Exclusion criteria: participation in work at any time; Individuals who have missed the modules and do not do the replacement later. Instruments: World Health Organization Quality of Life - (WHOQOL-BREF). Stress Perception Scale 10 (EPS-10) The Trait-State Anxiety Inventory: STAI E and T.

DETAILED DESCRIPTION:
INTRODUCTION - Personality is the set of characteristics that define the individual's behavior, his relationship with the external world and his way of reacting to the events that occur in it. Personality is closely related to the development of pathological processes, the integrity of your biological tissues and the repercussions that this can cause in your lives. In addition, there is a relationship with levels of anxiety, stress and quality of life. The enneagram is a tool that groups personalities into nine types, identifies their functioning patterns and reaction mechanisms. The use is quite widespread today, but still in an empirical way, requiring a greater scientific basis. OBJECTIVE - to observe the influence of the enneagram typology on the perception of anxiety, stress and quality of life through self-knowledge directed in a virtual learning environment. METHODS: clinical, primary, analytical, prospective and longitudinal study. It will be carried out in a virtual learning environment (VLE) with the collection of data obtained before and after the beginning of the training on the enneagram. The training will be divided into three online AVA modules. Casuistry: after orientations and signature of the term (Informed Consent Form), they will register on social networks where the initial information will be filled out. to outline the group. Inclusion criteria: participants of both sexes, Brazilians, over 18 years old; agree to sign the Informed Consent Form; with the desire to realize self-knowledge with the availability of time and access to the internet to hold meetings; Non-inclusion criteria: do not have previous information about the enneagram and speak the Portuguese language; Exclusion criteria: participation in work at any time; Individuals who have missed the modules and do not do the replacement later. Instruments: World Health Organization Quality of Life - (WHOQOL-BREF). Stress Perception Scale 10 (EPS-10) The Trait-State Anxiety Inventory: STAI E and T. After the guidance and signature of the ICF, the Organizational Learning Structure will be presented Statistical Analysis: The data will be tabulated in Microsoft Excel 2016 and measures will be used central tendency for quantitative variables and absolute and relative frequency for categorical variables. Pearson's correlation analysis; multiple regression analysis and Wilcoxon test. The product resulting from this work will be the Enneagram Online Teaching and Research System (Sep9). KEYWORDS: Personality. Anxiety. Quality of Life. Stress, Psychological. Personality Tests.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, Brazilians, adults, over 18 years old.
* Individuals who accept to sign the Informed Consent Form;
* Individuals with a desire to achieve self-awareness with the availability of time and access to the internet to hold meetings;

Exclusion Criteria:

* Individuals who drop out of work at any time;
* Individuals who have missed the modules and do not make a subsequent replacement;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Analysis of the condition of anxiety, stress and quality of life of the participating individuals. | Up to 24 weeks
  The data it will be tabulated in Microsoft Excel 2016 and submitted to statistical analysis, measures of central tendency were used for quantitative variables and absolute and relative frequency for categorical variables. The Minitabversion 18.1 program and the Statistical Package for the Social Sciences, Inc. (SPSS) Chicago, USA, version 22.0, were used. The level of significance used as a criterion for acceptance or rejection in the statistical tests was 5% (p <0.05).

SECONDARY OUTCOMES:
Analysis of the condition of anxiety, stress and quality of life of the participating after intervention with a virtual enneagram; . | through study completion, an average of 6 months
  The data were tabulated in Microsoft Excel 2016 and submitted to statistical analysis, measures of central tendency were used for quantitative variables and absolute and relative frequency for categorical variables. The Minitabversion 18.1 program and the Statistical Package for the Social Sciences, Inc. (SPSS) Chicago, USA, version 22.0, were used. The level of significance used as a criterion for acceptance or rejection in the statistical tests was 5% (p <0.05).

OTHER OUTCOMES:
Perception of self-knowledge after study and training through the virtual enneagram | through study completion, an average of 6 months
  The data were tabulated in Microsoft Excel 2016 and submitted to statistical analysis, measures of central tendency were used for quantitative variables and absolute and relative frequency for categorical variables. The Minitabversion 18.1 program and the Statistical Package for the Social Sciences, Inc. (SPSS) Chicago, USA, version 22.0, were used. The level of significance used as a criterion for acceptance or rejection in the statistical tests was 5% (p <0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Univás, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be available for download on the teaching platform.